CLINICAL TRIAL: NCT06903832
Title: Discharge Recommendations for Older Adults Using Physical Outcome Measure (DROP)
Brief Title: Discharge Recommendations for Older Adults Using Physical Outcome Measure
Acronym: DROP
Status: Recruiting | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/3331
Record Dates: First submitted 2025-03-28; First posted 2025-04-01 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Discharge Planning; Older Adults (65 Years and Older); Acute Hospitalization; OUTCOME MEASURES
Keywords: Discharge planning; Acute Hospitalization; Physical outcome measure; older adults; Gait Speed Test; Five Times Sit to Stand Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to explore if the use of Sit to Stand Test and Gait speed Test could assist physiotherapist with discharge planning decisions for older adults who are admitted to an acute hospital.

DETAILED DESCRIPTION:
Older adults are susceptible to acute illnesses which could predispose them to hospital admissions, with some of the common reasons for admission being infections, exacerbations of chronic conditions, and falls. This higher likelihood of older adults admitted to hospitals can be seen from the statistics from Ministry of Health in 2021 whereby older adults aged 65 years and older constitute up to 287.3 admissions per 1000 resident population, which is the highest among all age groups. In a study exploring the trend of injuries sustained by older adults presented to the Emergency Department of an acute hospital, 85.3% of all injuries sustained by older adults were due to falls. Common physical injuries sustained by older adults after a fall are fractures, bruises, and soft tissue injuries. Functional decline after a fall was also relatively common in older adults. Additionally, it has also been well recognized that hospitalisation may cause older adults to experience deconditioning. Therefore, older adults who are admitted to an acute hospital, especially those who are admitted due to falls or have a history of falls, are generally at high risk of having a change in their functional status. For the older adults with a change in functional status and have been assisted by a caregiver prior to their hospital admission, one of the main aims usually would be to make sure that their caregivers are still competent in caring for them after discharge. However, for older adults whose premorbid physical functional status are relatively independent, it is pertinent to establish if they are still safe to manage their own care after discharge from hospital. Proper discharge planning for this group of older adults is important to make sure that those who are discharge home will not experience functional decline or at increased risk of falls. Older adults who are admitted in an acute hospital are commonly referred to physiotherapists for assessment to determine are ready to return home or if they need further rehabilitation. However, to manage high workload in the acute hospital and space constraints in the wards, these older adults' readiness for home are frequently based on physiotherapists' clinical judgement, which may differ based on their clinical experience. Discharge planning is predominantly based on the comparisons between the older adults' self-reported functional mobility before hospital admission and the level of assistance they require during assessment by inpatient physiotherapists. Without the use objective outcome measures, there may be disagreement by medical team or family members on physiotherapist's recommendations. Furthermore, there is no venue to track the older adult's improvement objectively. STS and GST are two functional outcome measures that are validated to measure different physical aspects of older adults. STS has been shown to be able to assess lower limb strength, balance control and falls risk. This can be seen from the recommended use of STS in the acute setting for the assessment of lower limb strength and physical performance by a Singapore multidisciplinary consensus recommendation on muscle health in older adults by Chew et al. (2021). As for GST, it is reflective of a person's functional mobility whereby a study by Ostir et al., (2015) has demonstrated that GST can be used as a simple and quick screening tool for hospitalised older adults who may require further intervention with their mobility. As these two measures are easy to administer, less time-consuming and do not require much space, they may be suitable outcome measures to facilitate discharge planning. However, there is no literature demonstrating that they have been used to facilitate discharge planning for older adults in acute hospitals. Therefore, the primary aim of this study is to explore if the two outcome measures are useful in facilitating discharge planning for older adults who are admitted to an acute hospital. Our secondary aim is to determine if the discharge recommendations for participants to discharge home are accurate by looking for any change in the basic activity of living (ADL), self-reported fear of falls and activity confidence post-discharge

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and older
* Able to ambulate without physical assistance with or without walking aids as per premorbid status for at least 5 metres
* Clinical Frailty Scale (CFS) of ≤ 5
* Able to follow instructions (Abbreviated Mental Test (AMT) ≥ 5)

Exclusion Criteria:

* Admitted for acute orthopaedic or neurological conditions with physical deficits that affect functional mobility
* Requires physical assistance for functional mobility from ≥ 1 person
* Clinical Frailty Scale (CFS) of > 5
* AMT < 5 (Lack capacity to consent to study)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults admitted to inpatient wards in the National University Hospital (Singapore).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Five Times Sit To Stand Test (STS) | During Enrollment while admitted in acute hospital
  STS will be used to test the lower limb strength, balance control and falls risk. Participants will have to stand up and sit down five times started from a seated position, with arms across their chest. The test will have to be conducted as fast as possible using a chair with a backrest. The time taken to complete 5 repetitions will be recorded. Two trials will be performed. A cut-off score of ≥ 12s will be considered at risk of falling.
Gait Speed Test | During Enrollment while admitted in acute hospital
  A 4m walk test will be used to measure gait speed. Participant will walk through a 4-metre distance at comfortable speed. The time taken to complete the distance will be recorded. Two trials will be performed. Gait speed of ≤ 0.6m/s would be termed as dismobility according to Cummings et al., (2014) which would be reflected of having poor mobility and will require intervention.

SECONDARY OUTCOMES:
Calf Circumference | During Enrollment while admitted in acute hospital
  Calf circumference is a surrogate marker of muscle mass for older adults. It can be measured in sitting with the knee and ankle bent at a right angle and the feet flat on the floor. Using a measuring tape, the widest part of the part can be measured by applying the tape flat on the skin and parallel to the floor. Two measurements will be performed. A cut- off score of < 34cm in men and < 33cm in women will be consider as having low muscle mass and a higher risk of sarcopenia.
Hand grip strength | During Enrollment while admitted in acute hospital
  Hand grip strength measured by a hand dynamometer will be used to gauge frailty. Participant will sit in a chair with back support and asked to hold on to the dynamometer using maximum strength with the shoulder adducted and neutrally rotated, elbow flexed at 90 degrees, forearm neutral. The tested arm is not supported by examiner or armrest and the dynamometer is presented vertically and in line with the forearm. Three measurements will be performed. A cut off score of < 28kg in male and < 18kg in female is considered as having low handgrip strength.
Lower limb muscle strength using hand-held dynamometer | During Enrollment while admitted in acute hospital
  Reduction in quadriceps muscles strength were the most affected with aging. Muscle strength of lower limb will be assessed with knee extension strength using an electronic push/pull dynamometer. Participants would be seated with knee flexed to 90 degrees. Isometric knee strength will be measured with an electronic dynamometer attached to lower leg. A cut off score of < 23.64kg in male and < 15.24kg in female is considered as having low knee extension strength.
Modified Barthel Index (MBI) | During Enrollment while admitted in acute hospital and 2 weeks post-discharge
  The modified barthel index (MBI) consist of 10 items of ADLS modified from Barthel index (Shah et al, 1989). This includes transfers, walking, navigating stairs, grooming, bathing, dressing, feeding, toilet transfer, bladder and bowel control. It has been validated for older adults living at home and hospitalised older adults. MBI is also commonly used to assess physical function for hospitalised older adults at admission and discharge. MBI is positively associated with functional performance even for older adults who are hospitalised. In addition, older adults with higher MBI scores and ADL independence were more likely to be discharged home post hospitalisation as well. MBI score of 0 to 24 points suggest total ADL dependency, score of 25 to 49 points suggest severe ADL dependency, score of 50 to 74 suggest moderate ADL dependency and scores above 75 suggest mild ADL dependency.
Short Falls Efficacy Scale International (Short FES-I) | During Enrollment while admitted in acute hospital and 2 weeks post-discharge
  The Short FES-I measures the individual's concerns about falling. Seven questions were answered with a four-grade scale (1-4) of 'not at all concerned,' 'somewhat concerned,' 'fairly concerned' and 'very concerned.' The total score, which ranged from 7 to 28, was recorded. A higher score reflected a greater level of concern about falling. The Short FES-I have excellent psychometric properties and requires less time to conduct compared to the FES-I.
Balance Recovery Confidence scale (BRC) | During Enrollment while admitted in acute hospital and 2 weeks post-discharge
  The BRC aims to measure the balance recovery confidence in community-dwelling older adults. A list of fall-related situations commonly experienced by older adults are presented to determine how certain the respondent can recover their balance to prevent a fall if the situation was to occur in the last three weeks by recording a number from 0 to 10 with 10 indicating "Highly certain can do" and 0 refers to "Cannot do at all".
Mulitdimensional Falls Efficacy Scale (MdFES) | During Enrollment while admitted in acute hospital and 2 weeks post-discharge
  The MdFES was developed in collaboration between NUH and SIT (ITO Ref 2024-0720). The 4-item scale measures the perceived ability to prevent and manage falls. Participants will report their confidence levels on four items: (1) "How confident are you to walk steadily?"; (2) "How confident are you to stop yourself from falling when you lose balance?"; (3) "How confident are you to protect yourself if you fall?"; and (4) "How confident are you in getting up (from the ground) after a fall?" using a 5-point rating scale from 0 for "not at all confident" to 4 "Extremely confident". The scale has a high face and content validity and good internal consistency (α = .84).
Activities Balance Confidence scale (ABC) | During Enrollment while admitted in acute hospital and 2 weeks post-discharge
  The ABC scale assesses older adults' confidence that they will not fall or lose their balance when performing several progressively challenging balance and mobility tasks. This scale provides a broad continuum of activity difficulty and contains situation-specific questions to determine the level of confidence in completing a task without falling or losing balance. The ABC Scale has 16 items, with answers ranging from 0% (no confidence) to 100% (complete confidence)
Physical Activity Scale for the Elderly (PASE) | During Enrollment while admitted in acute hospital and 2 weeks post-discharge
  The PASE measures the level of self-reported physical activity in individuals aged 65 years or older. The scale has 12 items regarding occupational, household, and leisure activities during the previous 7-day period. The overall PASE score ranges from 0 to 400 or more with a higher score indicating greater level of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perera S, Mody SH, Woodman RC, Studenski SA. Meaningful change and responsiveness in common physical performance measures in older adults. J Am Geriatr Soc. 2006 May;54(5):743-9. doi: 10.1111/j.1532-5415.2006.00701.x. PMID 16696738
- [Result] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031
- [Result] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Result] Soh SLH, Ting HXT, Ho JY, Tan SL, Kayambu G, Koh KCGK, Low LL, Tan CYF. Assessing Falls Efficacy in Seniors: Important Insights in Hospital and Community Settings. J Frailty Sarcopenia Falls. 2025 Mar 1;10(1):48-53. doi: 10.22540/JFSF-10-048. eCollection 2025 Mar. PMID 40035087
- [Result] Soh SL, Tan CW, Xu T, Yeh TT, Bte Abdul Rahman F, Soon B, Gleeson N, Lane J. The Balance Recovery Confidence (BRC) Scale. Physiother Theory Pract. 2024 Mar 3;40(3):658-669. doi: 10.1080/09593985.2022.2135420. Epub 2022 Oct 19. PMID 36259660
- [Result] Kempen GI, Yardley L, van Haastregt JC, Zijlstra GA, Beyer N, Hauer K, Todd C. The Short FES-I: a shortened version of the falls efficacy scale-international to assess fear of falling. Age Ageing. 2008 Jan;37(1):45-50. doi: 10.1093/ageing/afm157. Epub 2007 Nov 20. PMID 18032400
- [Result] Shah S, Muncer S. Sensitivity of Shah, Vanclay and Cooper's modified Barthel Index. Clin Rehabil. 2000 Oct;14(5):551-2. doi: 10.1191/0269215500cr360oa. No abstract available. PMID 11043883
- [Result] Hang JA, Francis-Coad J, Naseri C, Jacques A, Waldron N, Purslowe K, Hill AM. Identifying the Association Between Older Adults' Characteristics and Their Health-Related Outcomes in a Transition Care Setting: A Retrospective Audit. Front Public Health. 2021 Jun 28;9:688640. doi: 10.3389/fpubh.2021.688640. eCollection 2021. PMID 34307282
- [Result] Pournajaf S, Pellicciari L, Proietti S, Agostini F, Gabbani D, Goffredo M, Damiani C, Franceschini M. Which items of the modified Barthel Index can predict functional independence at discharge from inpatient rehabilitation? A secondary analysis retrospective cohort study. Int J Rehabil Res. 2023 Sep 1;46(3):230-237. doi: 10.1097/MRR.0000000000000584. Epub 2023 Jun 16. PMID 37334818
- [Result] Aminalroaya R, Mirzadeh FS, Heidari K, Alizadeh-Khoei M, Sharifi F, Effatpanah M, Angooti-Oshnari L, Fadaee S, Saghebi H, Hormozi S. The Validation Study of Both the Modified Barthel and Barthel Index, and Their Comparison Based on Rasch Analysis in the Hospitalized Acute Stroke Elderly. Int J Aging Hum Dev. 2021 Oct;93(3):864-880. doi: 10.1177/0091415020981775. Epub 2020 Dec 18. PMID 33336587
- [Result] Ohura T, Hase K, Nakajima Y, Nakayama T. Validity and reliability of a performance evaluation tool based on the modified Barthel Index for stroke patients. BMC Med Res Methodol. 2017 Aug 25;17(1):131. doi: 10.1186/s12874-017-0409-2. PMID 28841846
- [Result] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Result] Menant JC, Weber F, Lo J, Sturnieks DL, Close JC, Sachdev PS, Brodaty H, Lord SR. Strength measures are better than muscle mass measures in predicting health-related outcomes in older people: time to abandon the term sarcopenia? Osteoporos Int. 2017 Jan;28(1):59-70. doi: 10.1007/s00198-016-3691-7. Epub 2016 Jul 9. PMID 27394415
- [Result] Abdalla PP, Dos Santos Carvalho A, Dos Santos AP, Venturini ACR, Alves TC, Mota J, de Sousa Oliveira A, Ramos NC, Marini JAG, Machado DRL. Cut-off points of knee extension strength allometrically adjusted to identify sarcopenia risk in older adults: A cross-sectional study. Arch Gerontol Geriatr. 2020 Jul-Aug;89:104100. doi: 10.1016/j.archger.2020.104100. Epub 2020 May 12. PMID 32470897
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Result] Rose Berlin Piodena-Aportadera M, Lau S, Chew J, Lim JP, Ismail NH, Ding YY, Lim WS. Calf Circumference Measurement Protocols for Sarcopenia Screening: Differences in Agreement, Convergent Validity and Diagnostic Performance. Ann Geriatr Med Res. 2022 Sep;26(3):215-224. doi: 10.4235/agmr.22.0057. Epub 2022 Aug 29. PMID 36031936
- [Result] Cummings SR, Studenski S, Ferrucci L. A diagnosis of dismobility--giving mobility clinical visibility: a Mobility Working Group recommendation. JAMA. 2014 May;311(20):2061-2. doi: 10.1001/jama.2014.3033. No abstract available. PMID 24763978
- [Result] Peters DM, Fritz SL, Krotish DE. Assessing the reliability and validity of a shorter walk test compared with the 10-Meter Walk Test for measurements of gait speed in healthy, older adults. J Geriatr Phys Ther. 2013 Jan-Mar;36(1):24-30. doi: 10.1519/JPT.0b013e318248e20d. PMID 22415358
- [Result] Ostir GV, Berges IM, Ottenbacher KJ, Fisher SR, Barr E, Hebel JR, Guralnik JM. Gait Speed and Dismobility in Older Adults. Arch Phys Med Rehabil. 2015 Sep;96(9):1641-5. doi: 10.1016/j.apmr.2015.05.017. Epub 2015 Jun 9. PMID 26067366
- [Result] Chew STH, Kayambu G, Lew CCH, Ng TP, Ong F, Tan J, Tan NC, Tham SL. Singapore multidisciplinary consensus recommendations on muscle health in older adults: assessment and multimodal targeted intervention across the continuum of care. BMC Geriatr. 2021 May 17;21(1):314. doi: 10.1186/s12877-021-02240-8. PMID 34001023
- [Result] Rydwik E, Bergland A, Forsen L, Frandin K. Investigation into the reliability and validity of the measurement of elderly people's clinical walking speed: a systematic review. Physiother Theory Pract. 2012 Apr;28(3):238-56. doi: 10.3109/09593985.2011.601804. Epub 2011 Sep 19. PMID 21929322
- [Result] Kim HJ, Park I, Lee HJ, Lee O. The reliability and validity of gait speed with different walking pace and distances against general health, physical function, and chronic disease in aged adults. J Exerc Nutrition Biochem. 2016 Sep;20(3):46-50. doi: 10.20463/jenb.2016.09.20.3.7. Epub 2016 Sep 30. PMID 27757387
- [Result] Goldberg A, Chavis M, Watkins J, Wilson T. The five-times-sit-to-stand test: validity, reliability and detectable change in older females. Aging Clin Exp Res. 2012 Aug;24(4):339-44. doi: 10.1007/BF03325265. PMID 23238309
- [Result] Chen Y, Almirall-Sanchez A, Mockler D, Adrion E, Dominguez-Vivero C, Romero-Ortuno R. Hospital-associated deconditioning: Not only physical, but also cognitive. Int J Geriatr Psychiatry. 2022 Mar;37(3):10.1002/gps.5687. doi: 10.1002/gps.5687. PMID 35142397
- [Result] Hoogerduijn JG, Buurman BM, Korevaar JC, Grobbee DE, de Rooij SE, Schuurmans MJ. The prediction of functional decline in older hospitalised patients. Age Ageing. 2012 May;41(3):381-7. doi: 10.1093/ageing/afs015. Epub 2012 Feb 28. PMID 22378613
- [Result] Loyd C, Markland AD, Zhang Y, Fowler M, Harper S, Wright NC, Carter CS, Buford TW, Smith CH, Kennedy R, Brown CJ. Prevalence of Hospital-Associated Disability in Older Adults: A Meta-analysis. J Am Med Dir Assoc. 2020 Apr;21(4):455-461.e5. doi: 10.1016/j.jamda.2019.09.015. Epub 2019 Nov 14. PMID 31734122
- [Result] Yeo YY, Lee SK, Lim CY, Quek LS, Ooi SB. A review of elderly injuries seen in a Singapore emergency department. Singapore Med J. 2009 Mar;50(3):278-83. PMID 19352571
- [Result] Zisberg A, Shadmi E, Gur-Yaish N, Tonkikh O, Sinoff G. Hospital-associated functional decline: the role of hospitalization processes beyond individual risk factors. J Am Geriatr Soc. 2015 Jan;63(1):55-62. doi: 10.1111/jgs.13193. PMID 25597557